CLINICAL TRIAL: NCT04816890
Title: A Phase 2 Trial to Assess the Efficacy and Safety of M1 Pram P037 Prandial Insulin in T1DM Subjects
Brief Title: A Trial to Assess the Efficacy and Safety of M1 Pram P037 Prandial Insulin in Subjects With Type 1 Diabetes (T1DM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adocia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT041-ADO09
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M1 Pram P037 (Experimental): Multi daily administration of M1 Pram P037 by subcutaneous injection
  Interventions: Drug: M1 Pram P037
- Insulin lispro (Active Comparator): Multi daily administration of insulin lispro (Humalog®) by subcutaneous injection
  Interventions: Drug: Insulin lispro

INTERVENTIONS:
Drug: M1 Pram P037 — Subcutaneous administration of M1 Pram P037 in combination with a basal insulin.
  Arms: M1 Pram P037
Drug: Insulin lispro — Subcutaneous administration of insulin lispro in combination with a basal insulin.
  Arms: Insulin lispro

SUMMARY:
In this trial, the treatment of subjects with type 1 diabetes with M1 Pram P037 as co-formulation of pramlintide and A21G human insulin analogue product will be compared with a current standard treatment, insulin lispro. During a four months treatment period doses in both treatment arms may be adjusted and optimised under outpatient conditions to allow a meaningful comparison of both treatments with respect to their effects on body weight, achievable glycaemic control, safety and tolerability, treatment satisfaction and well-being.

DETAILED DESCRIPTION:
After a run in period in case of basal insulin switch or Continuous Glucose Monitoring (CGM) initiation, eligible subjects will enter a 3 weeks baseline recording period.

Subjects will then be randomized to either M1 Pram P037 treatment or active comparator treatment (insulin lispro). Both investigator and enrolled subjects will be unblinded to treatment. Study participants will use CGM until follow-up visit.

Treatment period will last 16 weeks. Throughout the 4-month treatment period, basal insulin and investigational products administration will be individually adjusted. Treatment Satisfaction Questionnaire and WHO-5 well-being index will be completed by subjects at day 0 and after 2 months (Visit 9) and 4 months (Visit 11) of treatment.

A safety follow-up visit, 7 to 14 days after the last administration of IMP, will mark the end of the clinical trial for the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent obtained before any trial-related activities. Trial-related activities are any procedures that would not have been done during normal management of the subject.
* Subjects with type 1 diabetes mellitus.
* Body Mass Index (BMI) between 25.0 and 35.0 kg/m^2, both inclusive.
* HbA1c between 7.0 % and 9.5 %, both inclusive.
* Diabetes duration of at least 12 months.
* Using a multiple dosing insulin therapy (MDI) with a basal insulin and a rapid-acting insulin at at least two meals per day.
* Using any CGM or Flash Glucose Monitoring (FGM) for at least 1 month or willing to use CGM during the trial.

Exclusion Criteria:

* Known or suspected hypersensitivity to IMPs or any of the excipients or to any component of the IMP formulation.
* Type 2 diabetes mellitus.
* Receipt of any medicinal product in clinical development within 3 months or at least 5 half-lives of the related substances and their metabolites (whichever is longer) before randomisation in this trial.
* History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
* Any history or presence of cancer except basal cell skin cancer or squamous cell skin cancer as judged by the Investigator.
* Clinically significant abnormal screening laboratory tests, as judged by the Investigator.
* Systolic blood pressure < 90 mmHg or >139 mmHg and/or diastolic blood pressure < 50 mmHg or > 89 mmHg. One repeat test (on a different day, if necessary) will be acceptable in case of suspected white-coat hypertension.
* Clinically significant abnormal standard 12-lead electrocardiogram (ECG) after 5 minutes resting in supine position at screening, as judged by the Investigator.
* Proliferative retinopathy or maculopathy as judged by the Investigator based on a recent (<1.5 years) ophthalmologic examination.
* Severe neuropathy, in particular autonomic neuropathy, as judged by the Investigator.
* More than one episode of severe hypoglycaemia with seizure, coma or requiring assistance of another person during the past 6 months.
* Hypoglycaemic unawareness as judged by the Investigator.
* Hospitalisation for diabetic ketoacidosis during the previous 6 months.
* Presence of clinically significant gastrointestinal symptoms (e.g., nausea, vomiting, heartburn or diarrhea), as judged by the Investigator.
* Confirmed diagnosis of gastroparesis or requiring the use of drugs that alter gastrointestinal motility.
* Unusual meal habits and special diet requirements that could constitute a risk for the subject when participating in the trial or interfere with the interpretation of data.
* Use of oral antidiabetic drugs (OADs) and/or GLP-1 receptor agonists within 4 weeks prior to screening.
* Use of systemic glucocorticoid therapy (excluding topical, intraocular, intranasal, intra-articular, or inhaled preparations) within 2 months prior to screening.
* Use or planned use of drugs that promote weight loss (e.g. liraglutide, semaglutide, orlistat, lorcaserin, phentermine) within 2 months prior to screening.
* If female, pregnancy or breast-feeding.
* Women of childbearing potential who are not using a highly effective contraceptive method.
* The Investigator considers a subject as unsuitable for inclusion in the study for any other reason.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Body weight change from baseline to week 16 of treatment | From week 0 to week 16
  Change in body weight after 16 weeks of treatment

SECONDARY OUTCOMES:
TIR [70-180] mg/dL. | From week 0 to week 16
  Time In Range [70-180] mg/dL change from baseline to week 16 of treatment as measured by CGM.
%TIR [70-180] mg/dL. | From week 0 to week 16
  Percentage of Time In Range [70-180] mg/dL change from baseline to week 16 of treatment as measured by CGM.
TIR [70-140] mg/dL. | From week 0 to week 16
  Time In Range [70-140] mg/dL change from baseline to week 16 of treatment as measured by CGM.
%TIR [70-140] mg/dL. | From week 0 to week 16
  Percentage of Time In Range [70-140] mg/dL change from baseline to week 16 of treatment as measured by CGM.
MeanG_24h | From week 0 to week 16
  Average glucose over 24h change from baseline to week 16 of treatment
CVG_24h | From week 0 to week 16
  Coefficient Of Variation of glucose over 24h change from baseline to week 16 of treatment.
DistG_24h | From week 0 to week 16
  Distance travelled over 24h change from baseline to week 16 of treatment
SDG_24h | From week 0 to week 16
  Standard Deviation of all glucose values over 24h change from baseline to week 16 of treatment
HbA1c | From week 0 to week 16
  HbA1c change from baseline to week 16 of treatment
Total Insulin doses | From week 0 to week 16
  Change from baseline of total insulin doses
Prandial Insulin doses | From week 0 to week 16
  Change from baseline of prandial (per meal), insulin doses
Basal Insulin doses | From week 0 to week 16
  Change from baseline of basal insulin doses
Number of Adverse Events | From week 0 to week 16
  Number of Adverse Events observed during the treatment period
Duration of Adverse Events | From week 0 to week 16
  Duration of Adverse Events observed during the treatment period
Hypoglycaemic episodes | From week 0 to week 16
  Number of Hypoglycemic episodes during the 16 weeks treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Grit Andersen, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH; Eugen Baumgaertner, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (2):
- Germany (2):
  - Profil Mainz GmbH & Co, Mainz
  - Profil Institut für Stoffwechselforschung GmbH, Neuss

IPD SHARING:
Plan to Share IPD: No